CLINICAL TRIAL: NCT04187196
Title: Comparison of Bolus Dosing of Methohexital and Propofol in Elective Direct Current Cardioversion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00061732
Record Dates: First submitted 2019-11-26; First posted 2019-12-05 (Actual); Results first posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2021-11

CONDITIONS: Atrial Fibrillation; Atrial Flutter
Keywords: Cardioversion; Propofol; Deep sedation; Intravenous anesthetics
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter | interventions — Propofol; Methohexital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sedation with propofol group (Experimental): Participants in this group will be randomized to sedation with bolus dosing of propofol for cardioversion.
  Interventions: Drug: Propofol
- Sedation with methohexital group (Experimental): Participants in this group will be randomized to sedation with bolus dosing of methohexital for cardioversion.
  Interventions: Drug: Methohexital

INTERVENTIONS:
Drug: Propofol — Propofol will be given at an initial dose of 0.8 mg/kg followed by 20 mg every minute after 2 minutes, if adequate sedation is not achieved
  Other Names: Diprivan
  Arms: Sedation with propofol group
Drug: Methohexital — Methohexital will be given at an initial dose of 0.5 mg/kg, followed by 10 mg every minute after 2 minutes, if adequate sedation is not achieved
  Other Names: Brevital; Brietal
  Arms: Sedation with methohexital group

SUMMARY:
A randomized, open-blinded, prospective study to evaluate the timeliness and safety of direct current cardioversion (DCCV) when using methohexital when compared to the more often used propofol.

DETAILED DESCRIPTION:
The investigators theorize that the use of methohexital during cardioversion will result in a shorter time to effective sedation and time to full recovery when compared to the use of propofol. This will change how sedation is approached for elective cardioversions.

Primary Hypothesis:

1. The mean time to recovery from sedation during a cardioversion using methohexital for sedation will be significantly shorter than the recovery time using propofol for sedation, as evidenced by a short time from initiation of induction to a score of 2 on the Ramsay Sedation Scale.
2. The mean time to a Ramsay score of 5-6 will be significantly shorter using methohexital than the time to the same sedation level using propofol

Secondary Hypothesis:

1. There will be no significant increase in adverse events associated with the use of methohexital when compared with propofol.

ELIGIBILITY:
Inclusion Criteria:

* Patients who present to Wake Forest Baptist Medical Center for a direct current cardioversion for treatment of paroxysmal or persistent atrial fibrillation as well as atrial flutter.

Exclusion Criteria:

* Patients with sedation for transesophageal echocardiogram within 30 minutes of DCCV
* Hemodynamically compromised patients (as defined by hypotension <90/50 mmHg, altered mental status, shock, ischemic chest discomfort, or heart failure)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2020-04-29 (Actual); Primary Completion 2022-09-28 (Actual); Study Completion 2022-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elijah Beaty, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Medical Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Beaty EH, Fernando RJ, Jacobs ML, Winter GG, Bulla C, Singleton MJ, Patel NJ, Bradford NS, Bhave PD, Royster RL. Comparison of Bolus Dosing of Methohexital and Propofol in Elective Direct Current Cardioversion. J Am Heart Assoc. 2022 Oct 4;11(19):e026198. doi: 10.1161/JAHA.122.026198. Epub 2022 Sep 21. PMID 36129031

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sedation With Propofol Group | Sedation With Methohexital Group
Started | 35 | 38
Completed | 33 | 38
Not Completed | 2 | 0
Not completed — Screen Failure | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sedation With Propofol Group | Sedation With Methohexital Group | Total
Number analyzed (Participants) | 33 | 38 | 71
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 7 | 17
  >=65 years | 23 | 31 | 54
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 16 | 29
  Male | 20 | 22 | 42
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 5 | 8
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 30 | 33 | 63
Region of Enrollment [Number; unit: participants]
  United States | 33 | 38 | 71
Body Mass Index (BMI) [Median (Inter-Quartile Range); unit: kg/m^2] | 30.7 [26.1 to 36.6] | 30.8 [26.6 to 36.3] | 30.7 [26.3 to 36.4]
CHA2 DS2-VASc Congestive heart failure, Hypertension, Diabetes mellitus, prior Stroke [Median (Inter-Quartile Range); unit: score on a scale] — congestive heart failure, hypertension, age ≥75 (doubled), diabetes, stroke (doubled), vascular disease, age 65 to 74 and sex category (female)(CHA2 DS2-VASc ); a score of 0 is "low" risk of stroke, 1 is "moderate", and any score above 1 is a "high" risk - scores range from 0-4 with 4 meaning higher risk of stroke
  score on a scale | 3 [2 to 4.5] | 3 [2.8 to 5.0] | 3 [2 to 5]
HAS-BLED score (Hypertension, Abnormal renal/liver function, Stroke, Bleeding history [Median (Inter-Quartile Range); unit: score on a scale] — HAS-BLED is an acronym of the major factors associated with bleeding risk: Hypertension, Abnormal renal and liver function, Stroke, Bleeding, Labile International Normalized Ratio (INR), Elderly, Drugs or alcohol; The score predicts major bleeding risk. Score is between 0 and 9 score of ≥ 3 indicates a high risk of bleeding.
  score on a scale | 2 [1 to 3] | 2 [1 to 3] | 2 [1 to 3]
Left Atrium (LA) Diameter [Median (Inter-Quartile Range); unit: cm] | 4.3 [3.9 to 4.6] | 4.3 [3.8 to 5.2] | 4.3 [3.9 to 4.9]
Left Ventricle ejection fraction (LVEF) [Median (Inter-Quartile Range); unit: percentage of blood] — Ejection fraction refers to how well your heart pumps blood. It is the amount of blood pumped out of your heart's lower chambers (ventricles) each time it contracts. An ejection fraction in a healthy heart is 50% to 70%
  percentage of blood | 60 [55 to 60] | 60 [51 to 65] | 60 [55 to 65]
Number with History of Hypertension [Count of Participants; unit: Participants] | 29 | 34 | 63
History of heart failure with reduced ejection fraction (HFrEF) [Count of Participants; unit: Participants] | 3 | 8 | 11
History of Transient Ischemic attack (TIA) or stroke [Count of Participants; unit: Participants] | 4 | 3 | 7
Number with History of Diabetes [Count of Participants; unit: Participants] | 11 | 11 | 22
Number with History of Chronic Obstructive Pulmonary Disease (COPD) [Count of Participants; unit: Participants] | 6 | 6 | 12
Number with Thyroid Disorder [Count of Participants; unit: Participants] | 11 | 10 | 21
Number Currently Smoking [Count of Participants; unit: Participants] | 6 | 3 | 9
Number Drinking at Least 1 Time per Week [Count of Participants; unit: Participants] | 9 | 14 | 23
Number of Drinkers having >2 drinks per occasion [Count of Participants; unit: Participants] | 4 | 4 | 8
American Society of Anesthesiologists (ASA) classification III or IV [Count of Participants; unit: Participants] — ASA classification III--someone with severe systemic disease, Substantive functional limitations. ASA classification IV--someone with a severe systemic disease that is a constant threat to life.
  Participants | 26 | 32 | 58
Heart Rate [Median (Inter-Quartile Range); unit: beats per minute (bpm)] | 96 [79 to 115] | 93 [77 to 128] | 94 [78 to 118]
Systolic Blood Pressure [Median (Inter-Quartile Range); unit: mmHg] | 132 [125.5 to 146] | 140 [132 to 151.3] | 138 [128 to 151]
Diastolic Blood Pressure [Median (Inter-Quartile Range); unit: mmHg] | 78 [67.5 to 98.5] | 79.5 [71 to 93] | 79 [71 to 94]
Median arterial pressure [Mean (Inter-Quartile Range); unit: mmHg] | 104 [91 to 113] | 104.5 [96.5 to 118.3] | 104 [94 to 117]
Respiratory Rate [Median (Inter-Quartile Range); unit: respirations per minute (rpm)] | 16 [12.5 to 20] | 16.5 [14 to 21.3] | 16 [13 to 21]
Oxygen saturation % [Median (Inter-Quartile Range); unit: percentage of oxygen saturation] | 100 [99 to 100] | 100 [99 to 100] | 100 [99 to 100]

OUTCOME MEASURES:

1. Primary Outcome: Time From Initiation of Sedation to Full Recovery
Description: The time from initiation of sedation to full recovery Ramsay Sedation Scale (RSS) of 2 (RSS 2 means awake; cooperative, oriented, and tranquil.)-- as evidenced by the ability to answer the questions "What is your name and what is your age?" The timer will start at the initiation of induction. Recorded in minutes.
Time Frame: Day 1
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Sedation With Propofol Group | Sedation With Methohexital Group
Number analyzed (Participants) | 33 | 38
minutes | 7.6 [6.5 to 9.8] | 5.5 [4.0 to 6.9]

2. Secondary Outcome: Time From End of Injection to Loss of Conscious
Description: Recorded in minutes.
Time Frame: Day 1
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Sedation With Propofol Group | Sedation With Methohexital Group
Number analyzed (Participants) | 33 | 38
minutes | 1.0 [0.8 to 1.3] | 1.0 [0.8 to 1.3]

3. Secondary Outcome: Time to First Electrical Direct-current Shock
Description: Recorded in seconds.
Time Frame: Day 1
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Sedation With Propofol Group | Sedation With Methohexital Group
Number analyzed (Participants) | 33 | 38
seconds | 1.28 [0.8 to 3.3] | 1.2 [1.0 to 1.7]

4. Secondary Outcome: Time to Eyes Opening
Description: Recorded in seconds.
Time Frame: Day 1
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Sedation With Propofol Group | Sedation With Methohexital Group
Number analyzed (Participants) | 33 | 38
seconds | 7.0 [5.7 to 9.6] | 4.2 [3.3 to 6.4]

5. Secondary Outcome: Systolic Blood Pressure
Time Frame: Day 1: at induction, prior to first shock, and 1 minute, 3 minutes, 5 minutes, 7 minutes, 9 minutes, 10 minutes, 15 minutes, 20 minutes and 30 minutes after first cardioversion
Measure: Median (Inter-Quartile Range); unit: mmHg
Arm/Group | Sedation With Propofol Group | Sedation With Methohexital Group
Number analyzed (Participants) | 33 | 38
mmHg
  at induction | 132 [125.5 to 146] | 140 [132 to 151.3]
  prior to first shock | 138 [125 to 148] | 144 [130 to 153]
  1 minute after first cardioversion | 124 [107 to 139.5] | 132 [121.8 to 155.3]
  3 minutes after first cardioversion | 122 [106.5 to 131.5] | 140.5 [124 to 157.5]
  5 minutes after first cardioversion | 114 [106 to 126] | 142.5 [124.8 to 158.3]
  7 minutes after first cardioversion | 111 [101 to 122] | 139.5 [123.3 to 151]
  9 minutes after first cardioversion | 111 [96 to 129] | 131 [120 to 143.3]
  10 minutes after first cardioversion | 113 [94.5 to 123] | 136 [123.8 to 141.3]
  15 minutes after first cardioversion | 113 [99.3 to 122.8] | 131 [115.5 to 141.5]
  20 minutes after first cardioversion | 116 [101.3 to 127.8] | 127 [118 to 137]

6. Secondary Outcome: Diastolic Blood Pressure
Time Frame: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: mmHg
Arm/Group | Sedation With Propofol Group | Sedation With Methohexital Group
Number analyzed (Participants) | 33 | 38
mmHg
  at induction | 78 [67.5 to 98.5] | 79.5 [71 to 93]
  prior to first shock | 82 [69 to 96] | 81.5 [72 to 91.5]
  1 minute after first cardioversion | 70 [58.5 to 83.5] | 76 [67.8 to 89.3]
  3 minutes after first cardioversion | 65 [59.5 to 75.5] | 74 [66.8 to 82]
  5 minutes after first cardioversion | 65 [57 to 75.5] | 73 [69.3 to 79]
  7 minutes after first cardioversion | 63 [56.5 to 71] | 72 [66.5 to 78]
  9 minutes after first cardioversion | 60 [56 to 72.5] | 68 [63 to 74.3]
  10 minutes after first cardioversion | 67 [57 to 73] | 68 [63 to 74]
  15 minutes after first cardioversion | 65 [56.5 to 76.8] | 69 [62.5 to 74.5]
  20 minutes after first cardioversion | 66 [56.5 to 73] | 66 [61 to 76.5]
  30 minutes after first cardioversion | 67 [59.3 to 75.8] | 67 [61 to 73]

7. Secondary Outcome: Mean Arterial Blood Pressure
Time Frame: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: mmHg
Arm/Group | Sedation With Propofol Group | Sedation With Methohexital Group
Number analyzed (Participants) | 33 | 38
mmHg
  at induction | 104 [91 to 113] | 104.5 [96.5 to 118.3]
  prior to first shock | 102 [91.5 to 117.5] | 104.5 [92.8 to 115]
  1 minute after first cardioversion | 91 [74 to 104] | 101.5 [90.5 to 110]
  3 minutes after first cardioversion | 86 [80.5 to 96.5] | 104 [89.8 to 109.8]
  5 minutes after first cardioversion | 84 [78 to 96] | 101 [91 to 112.3]
  7 minutes after first cardioversion | 81 [72.5 to 91.5] | 99.5 [88 to 106.3]
  9 minutes after first cardioversion | 81 [72 to 93] | 95 [85.8 to 102]
  10 minutes after first cardioversion | 84 [72.5 to 92.5] | 94 [88.3 to 100]
  15 minutes after first cardioversion | 85 [76 to 92.8] | 92 [84.5 to 99]
  20 minutes after first cardioversion | 86 [75.3 to 91.5] | 92 [85 to 98]
  30 minutes after first cardioversion | 87 [78.8 to 106.1] | 93 [85.5 to 99.5]

8. Secondary Outcome: Respiratory Rate
Time Frame: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: number of breaths per minute
Arm/Group | Sedation With Propofol Group | Sedation With Methohexital Group
Number analyzed (Participants) | 33 | 38
number of breaths per minute
  at induction | 16 [12.5 to 20] | 16.5 [14 to 21.3]
  prior to first shock | 18 [13.5 to 21.5] | 16.5 [14.8 to 23]
  1 minute after first cardioversion | 17 [11 to 22] | 17 [12.8 to 22]
  3 minutes after first cardioversion | 19 [15 to 22.5] | 19.5 [17 to 22.3]
  5 minutes after first cardioversion | 19 [16 to 22.5] | 18.5 [16 to 22.3]
  7 minutes after first cardioversion | 19 [15.5 to 22] | 19.5 [15 to 22]
  9 minutes after first cardioversion | 18 [15.5 to 22.5] | 17 [15 to 21.5]
  10 minutes after first cardioversion | 18 [15.5 to 21.5] | 18 [13.5 to 22.3]
  15 minutes after first cardioversion | 18 [13 to 22] | 17 [15 to 20.5]
  20 minutes after first cardioversion | 17 [15 to 20] | 18 [15 to 21]
  30 minutes after first cardioversion | 18 [16 to 20] | 18 [15 to 20.5]

9. Secondary Outcome: Saturation of Peripheral Oxygen (SpO2)
Time Frame: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: percentage of oxygen saturation
Arm/Group | Sedation With Propofol Group | Sedation With Methohexital Group
Number analyzed (Participants) | 33 | 38
percentage of oxygen saturation
  at induction | 100 [99 to 100] | 100 [99 to 100]
  prior to first shock | 100 [99.5 to 100] | 100 [100 to 100]
  1 minute after first cardioversion | 98 [97 to 100] | 99.5 [97.8 to 100]
  3 minutes after first cardioversion | 99 [97.5 to 100] | 100 [98.8 to 100]
  5 minutes after first cardioversion | 99 [99 to 100] | 100 [99 to 100]
  7 minutes after first cardioversion | 99 [99 to 100] | 100 [99 to 100]
  9 minutes after first cardioversion | 100 [99 to 100] | 100 [99 to 100]
  10 minutes after first cardioversion | 100 [98 to 100] | 100 [98 to 100]
  15 minutes after first cardioversion | 100 [98 to 100] | 100 [98 to 100]
  20 minutes after first cardioversion | 99 [98 to 100] | 99 [98 to 100]
  30 minutes after first cardioversion | 98 [97 to 100] | 98 [96.5 to 99.5]

10. Secondary Outcome: Heart Rate
Time Frame: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: beats per minute
Arm/Group | Sedation With Propofol Group | Sedation With Methohexital Group
Number analyzed (Participants) | 33 | 38
beats per minute
  at induction | 96 [79 to 115] | 93 [77 to 128]
  prior to first shock | 100 [84.5 to 118.5] | 92 [75.8 to 122]
  1 minute after first cardioversion | 69 [62.5 to 78] | 73.5 [66 to 84.3]
  3 minutes after first cardioversion | 66 [60 to 76.5] | 73.5 [62.5 to 84.5]
  5 minutes after first cardioversion | 69 [61 to 74] | 69 [60.8 to 81.3]
  7 minutes after first cardioversion | 66 [59.5 to 71.5] | 69 [59.8 to 78.3]
  9 minutes after first cardioversion | 65 [59 to 73] | 67.5 [60.8 to 78.3]
  10 minutes after first cardioversion | 64 [58 to 74] | 68 [59.5 to 79.3]
  15 minutes after first cardioversion | 64.5 [59 to 72.5] | 68 [59.5 to 77.5]
  20 minutes after first cardioversion | 62.5 [58.3 to 72] | 68 [59.5 to 74.5]
  30 minutes after first cardioversion | 65.5 [61 to 72.3] | 69 [60 to 75.5]

11. Secondary Outcome: Recall of Pain at Injection Site - Visual Analog Scale
Description: These are 100 mm lines that are anchored with "no pain" on one end and "worst imaginable pain" on the other end. Total range 0-100, higher numbers correspond to worse pain.
Time Frame: Day 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Sedation With Propofol Group | Sedation With Methohexital Group
Number analyzed (Participants) | 33 | 38
score on a scale | 8 [1 to 46] | 2 [0 to 11.5]

12. Secondary Outcome: Recall of Anything Unpleasant About the Procedure - Visual Analog Scale
Description: These are 100 mm lines that are anchored with "no distress" on one end and "worst imaginable distress" on the other end. Total range 0-100, higher numbers correspond to worse distress.
Time Frame: Day 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Sedation With Propofol Group | Sedation With Methohexital Group
Number analyzed (Participants) | 33 | 38
score on a scale | 3 [0 to 19] | 1 [0 to 12.5]

ADVERSE EVENTS:
Time Frame: Baseline through the end of study (approximately 1 day)
Arm/Group | Sedation With Propofol Group | Sedation With Methohexital Group
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/38
Serious Adverse Events (participants affected / at risk) | 1/33 | 0/38
Other Adverse Events (participants affected / at risk) | 14/33 | 24/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sedation With Propofol Group (N=33) | Sedation With Methohexital Group (N=38)
Severe Oxygen Desaturation (<75% or <90% at 60s) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sedation With Propofol Group (N=33) | Sedation With Methohexital Group (N=38)
Bradycardia (Cardiac disorders) | 11 (12) | 12 (12)
Hypotension (Cardiac disorders) | 14 (14) | 4 (4)
Hypoxemia (Social circumstances) | 5 (5) | 0 (0)
Jaw thrust or chin lift (Musculoskeletal and connective tissue disorders) | 14 (14) | 6 (6)
Apnea >20 seconds (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-08-26): https://cdn.clinicaltrials.gov/large-docs/96/NCT04187196/Prot_SAP_000.pdf
  • Informed Consent Form (2020-12-09): https://cdn.clinicaltrials.gov/large-docs/96/NCT04187196/ICF_001.pdf